CLINICAL TRIAL: NCT06282614
Title: MOVHYDA (MUCO245) - Performance and Safety of MUCOGYNE® Ovule as a Moisturizer
Brief Title: Performance and Safety of MUCOGYNE® Ovule as a Moisturizer
Acronym: MOVHYDA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Early efficacy at interim analysis.
Sponsor: Biocodex (Industry)
Collaborators: Voisin Consulting Life Science (VCLS) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MUCO245; 2023-A02081-44 (Other: ID-RCB)
Record Dates: First submitted 2024-02-01; First posted 2024-02-28 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Vaginal Dryness

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter (France), open label without comparator study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mucogyne treatment (Experimental): 2 planned visits for each eligible patient :
  * Screening/Baseline visit : V1 at Day 0. Patient receive Mucogyne Ovule.
  * End-of-study visit : V2 at Day 35 ± 3
  Interventions: Device: Mucogyne Ovule

INTERVENTIONS:
Device: Mucogyne Ovule — At inclusion visit (V0), the Investigator will ask the subject to use MUCOGYNE® Ovule 2 times a week until symptoms improve during 5 weeks (D35± 3) preferably at bedtime

SUMMARY:
The aim of this post-Market Clinical Follow-up (PMCF) study is to confirm the efficacy and safety of MUCOGYNE® Ovule in the maintainance of natural moisture of the vulvovaginal mucosa and in the compensation for any natural secretions deficiencies, when used in accordance with its approved labeling, in the context of vulvovaginal dryness.

ELIGIBILITY:
Inclusion Criteria:

Women with the following conditions:

* ≥ 18 years of age at inclusion with vaginal dryness, irrespective of the cause (which may or may not be accompanied by irritation of the vulva, discomfort, or itchiness) : women who suffer pain during sexual intercourse, women taking the mini pill, mothers during breastfeeding, menopausal women and women taking anti-acne treatment.
* Having a Vaginal Health Index Score (VHIS) <15 associated to pain and/or dyspareunia feeling.
* If the patient has reproductive potential, she must be willing to use effective method of contraception (oral contraceptive, intrauterine device, subcutaneous contraceptive implant, vaginal ring, and condom).
* Patient agrees to not use any local oestrogens, or other vaginal product during the study
* Patient agrees to not modify their intimate hygiene and lubricant products
* Patient able to understand and sign the informed consent form before beginning any study procedure
* Patient able to comply with study requirements, as defined in the protocol.
* Patient affiliated to a health social security system.

Exclusion Criteria:

Women with the following conditions:

General criteria:

* Pregnant women (patient of childbearing potential must not be pregnant and must agree to avoid pregnancy during the study by using an effective birth control method from at least one month before D0 (V1) and throughout the duration of the study)
* Patient participating at the same time in another interventional trial within the four previous weeks and during the study period, being in an exclusion period for a previous study
* Patient deprived of freedom by administrative or legal decision or under guardianship
* Patient in a social or sanitary establishment
* Patient suspected to be non-compliant according to the investigator's judgment
* Patient in an emergency situation

Criteria related to patient's status:

* Patient with known hypersensitivity to one of MUCOGYNE® Ovule components
* Patient with a known vaginal pathology (clinical diagnosis only) other than vaginal dryness/atrophy

Criteria related to previous or ongoing treatments:

* Patient with a condition or receiving a medication which, in the investigator's judgment, put the patient at undue risk
* Patient suffering from systemic diseases and/or using concurrent therapy that may interfere with the evaluation of the study results
* Patient undergoing a topical treatment on the test area or a systemic treatment such as:

  * corticosteroids during the 2 previous weeks and during the study
  * retinoids and/or immunosuppressors during the 1.5 previous months and during the study
  * Patient having started or changed her oral contraceptive or any other hormonal treatment during the three previous months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 33 (Actual)
Dates: Start 2024-04-11 (Actual); Primary Completion 2025-02-14 (Actual); Study Completion 2025-02-14 (Actual)

PRIMARY OUTCOMES:
Assessment of the efficacy of MUCOGYNE® Ovule intra vaginal applications on subjects' vaginal dryness irrespective of the cause over a 35-day period of use | Day 0 to Day 35 ± 3
  Primary efficacy criterion: Clinical scoring, by the investigator, of the Vaginal Health Index Score (VHIS), including evaluation of elasticity, fluid volume, pH, epithelial integrity, and moisture. The minimum score is 5 and the maximum score is 25. If VHIS <15, the vagina is considered atrophic.

SECONDARY OUTCOMES:
Assessment of the local performance of MUCOGYNE® Ovule in reducing vulva irritation | Day 0 to Day 35 ± 3
  Secondary efficacy criteria : Auto-evaluation, by the subjects, of vulva irritation on Visual Analogical Scales (VAS) from 0 to 10
Assessment of the local performance of MUCOGYNE® Ovule in reducing vulvo-vaginal discomfort | Day 0 to Day 35 ± 3
  Secondary efficacy criteria : Auto-evaluation, by the subjects, of discomfort on Visual Analogical Scales (VAS) from 0 to 10
Assessment of the local performance of MUCOGYNE® Ovule in reducing itching | Day 0 to Day 35 ± 3
  Secondary efficacy criteria : Auto-evaluation, by the subjects, of itching on Visual Analogical Scales (VAS) from 0 to 10
Assessment of the local performance of MUCOGYNE® Ovule in reducing pain and/or dyspareunia related to vaginal dryness | Day 0 to Day 35 ± 3
  Secondary efficacy criteria : Auto-evaluation, by the subjects, of pain and/or dyspareunia on Visual Analogical Scales (VAS) from 0 to 10
Assessment of the patient's sexual function | Day 0 to Day 35 ± 3
  Secondary efficacy criteria : Completion of the self-reported FSFI (Female Sexual Function Index) to investigate sexual function (for women having sexual relations). The minimum score is 2 and the maximum score is 36. An alteration in sexuality is a score less than or equal to 26,55.
Assessment of the patient's satisfaction | Day 0 to Day 35 ± 3
  Secondary efficacy criteria :
  * Completion of the intra vaginal treatment satisfaction questionnaire (Likert questionnaire) to assess the level of satisfaction of the treatment on the vaginal symptoms. Two questions with 5 possible answers :
  * 1 : Strongly agree
  * 2 : Agree
  * 3 : Neither
  * 4 : Disagree
  * 5 : Strongly disagree
Assessment of changes in patient's clinical status | Day 0 to Day 35 ± 3
  Secondary efficacy criteria :Completion of the Patients' Global Impression of Change (PGIC) Scale to assess the changes perceived by the patient following the treatment taken from 1 to 7. An improvement is a score from 1 to 3 whereas a deterioration is a score of 5 to 7. A score of 4 means stability.
Assessment by investigator of changes in patient's clinical status | Day 0 to Day 35 ± 3
  Secondary efficacy criteria :Completion of the Clinical Global Impressions-Improvement (CGI-I) by the investigator to assess the changes following the treatment taken from 1 to 7. An improvement is a score from 1 to 3 whereas a deterioration is a score of 5 to 7. A score of 4 means stability.
Assessment of the safety of MUCOGYNE® Ovule | Day 0 to Day 35 ± 3
  Secondary efficacy criteria : Reporting of number, nature and characteristics of any adverse event : incidence, seriousness, severity, resolution.
Assessment of the device deficiencies of MUCOGYNE® Ovule | Day 0 to Day 35 ± 3
  Secondary efficacy criteria : Reporting of Device deficiencies: type of deficiency, batch number, action taken, consequence of deficiency.
Assessment of the usability of MUCOGYNE® Ovule | Day 0 to Day 35 ± 3
  Secondary efficacy criteria :
  * Completion of the usability question by the patient. There are 4 possible answers :
  * Very easy
  * Easy
  * Difficult
  * Very Difficult

CONTACTS AND LOCATIONS:
Overall Officials: Oana BERNARD, MD, Study Director — Chief Scientific Officer
Locations (3):
- France (3):
  - Dr Ramez GHADRI's medical office, Orléans, France
  - JEAN Christian's medical office, Nogent-sur-Marne
  - Dr Raïssa APERANO-MAS's medical office, Rennes

IPD SHARING:
Plan to Share IPD: No